CLINICAL TRIAL: NCT03511547
Title: Arthroscopic Rotator Cuff Reconstruction With or Without Biologic or Synthetic Patch Augmentation in Patients Over 60 Years: a Randomized Controlled Trial
Brief Title: Comparison of Arthroscopic Supraspinatus Tendon Tear Repair in Patients Over 60 Years With and Without Patch Augmentation.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Personal reasons
Sponsor: Schulthess Klinik (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARCR-RCT
Record Dates: First submitted 2018-04-18; First posted 2018-04-30 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2018-04

CONDITIONS: Rotator Cuff Tears
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention group 1: Pitch-Patch (Active Comparator): Reconstruction with patch augmentation using a synthetic patch
  Interventions: Device: Pitch Patch
- Intervention group 2: ArthroFlex (Active Comparator): Reconstruction with patch augmentation using a biological human dermis patch
  Interventions: Device: ArthroFlex
- Control (No Intervention)

INTERVENTIONS:
Device: Pitch Patch — The patients will be operated by shoulder arthroscopy according to the internationally standardized procedure. Patients allocated this group will receive a synthetic (Pitch-Patch™ [PP]) augmentation.
  Arms: Intervention group 1: Pitch-Patch
Device: ArthroFlex — The patients will be operated by shoulder arthroscopy according to the internationally standardized procedure. Patients allocated this group will receive a biologic patch (ArthroFlex® [AF]) augmentation.
  Arms: Intervention group 2: ArthroFlex

SUMMARY:
The aim of the study is to show that patch augmentation in rotatorcuff tear results in lower rate of recurrent tendon defects compared without patches.

DETAILED DESCRIPTION:
An arthroscopic rotator cuff repair is nowadays mostly implemented in order to restore function and reduce or eliminate pain. The primary objective of this randomized controlled trial is to demonstrate, in patients 60 years or older with a large rotator cuff tear, that biological or synthetic patch augmen-tation in arthroscopic rotator cuff repair results in decreased rate of retear 24 months post-operatively compared to re-pair without patch augmentation.

ELIGIBILITY:
Inclusion Criteria:

* Rotator cuff tear > 2 cm in the sagittal plane involving the supraspinatus tendon as well as at least the superior 1/3 of the infraspinatus tendon
* Indicated for surgical reconstruction by arthroscopy
* Patient aged 60 years and over
* Consenting participation in this study by signing the Informed Consent form

Exclusion Criteria:

* Osteoarthritis (grade ≥ 2 after Samilson & Prieto)
* Advanced fatty infiltration of the rotator cuff muscles (Goutallier grade III or IV)
* Tear of the subscapularis > Typ 1 Lafosse (partial tears of superior 1/3 of the tendon)
* Irreparable tear of the supraspinatus
* General medical contraindication to surgery
* Known hypersensitivity to the materials used
* Revision operations
* Open reconstruction
* Tendon transfer necessary (latissimus dorsi or pectoralis major)
* Any disease process that would preclude accurate evaluation including:

  * Systemic arthritis, rheumatoid arthritis, diabetes (insulin dependent), acute or chronic infection, abnormal bone metabolism, tumour / malignoma, psychiatric disorder
  * Inadequate blood flow or neuromuscular disease in the affected arm
* Recent history of substance abuse
* Legal incompetence
* German language barrier to complete the questionnaires or
* Participation in any other medical device or medicinal product study that could influence the results of the present study

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Occurrence of retear | 24 months
  Repair integrity will be assessed by an independent assessor on the basis of centralized MRI images.

SECONDARY OUTCOMES:
Pain level (NRS) | 6/24 months
  The pain level in the operated shoulder will be measured with a numeric rating scale (0=no pain, 10 = maximum pain) as part as the Constant Murley Score (CS)
Range of motion (flexion, abduction, external and internal rotation) | 6/24 months
  The following active and passive range of motion parameters of the affected shoulder will be documented using a goniometer : Elevation (flexion), abduction, External rotation by 0° abduction, external-internal rotation by 90° abduction
Shoulder strength in 90° abduction and in external rotation (0° abduction) | 6/24 months
  The shoulder strenght will be measured with an isobex device
Constant Murley Score (CS) | 6/24 months
  The CMS is a 100-point scoring system that is divided into four subscales: pain (15 points), activities of daily living (20 points), range of motion (40 points) and strength (25 points).Pain and activities of daily living are self-reported by the patient using visual analog scales and ordinal categories. Range of motion is obtained during active painfree elevation in flexion and abduction (using a goniometer), and functional internal and external rotation of the shoulder (using ordinal scale). Strength testing was performed at 90° of abduction in the scapular plane.
Oxford Shoulder Score (OSS) | 6/24 months
  The Oxford Shoulder Score used after 3 months is the primary parameter. The Score tests the ability to participate in the patients' normal life before they got injured.
Subjective shoulder value (SSV) | 6/24 months
  The Subjective Shoulder Value (SSV) is based on a single question that is answered subjectively by the patients. The English formulation of this question is: "What is the overall percent value of your shoulder if a completely normal shoulder represents 100%?"
Quality of life (utilities) and general health using EQ-5D-5L | 6/24 months
  EQ-5D is a standardised measure of health status developed by the EuroQol Group in order to provide a simple, generic measure of health for clinical and economic appraisal.Applicable to a wide range of health conditions and treatments, it provides a simple descriptive profile and a single index value for health status that can be used in the clinical and economic evaluation of health care as well as in population health surveys.
Subjective improvement, expectation, satisfaction with treatment | 6/24 months
  Patients will be asked to assess their current state of health related to the operated shoulder at follow-up compared to the state before surgery. Further on A similar question will be asked regarding their perceived change in quality of life.At the 24-month follow-up questionnaire, patients will rate whether the surgical results met their expectations:
Adverse events / complications | 3/6/24 months and intra-operative
  Adverse events will be analyzed according to their type and time of occurrence, severity and relation-to-implant: Local AEs within 24 months and Non-local AEs within 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Markus Scheibel, Prof, Principal Investigator — Schulthess Klinik

IPD SHARING:
Plan to Share IPD: No